CLINICAL TRIAL: NCT01042977
Title: A 24-week, Multicentre, Randomised, Double-blind,Age-stratified, Placebo Controlled Phase III Study With an 80-week Extension Period to Evaluate the Efficacy and Safety of Dapagliflozin 10 mg Once Daily in Patients With T2DM and Cardiovascular Disease, Who Exhibit Inadequate Glycaemic Control on Usual Care
Brief Title: Efficacy and Safety in Patients With Type 2 Diabetes Mellitus and Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D1690C00019
Record Dates: First submitted 2010-01-05; First posted 2010-01-06 (Estimated); Results first posted 2013-08-23 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2013-12

CONDITIONS: Type 2 Diabetes Mellitus; Cardiovascular Disease; Inadequate Glycaemic Control
Keywords: dapagliflozin; diabetes; cardiovascular disease
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Cardiovascular Diseases; Diabetes Mellitus | interventions — dapagliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): dapagliflozin 10 mg tablet
  Interventions: Drug: Dapagliflozin
- 2 (Placebo Comparator): matching placebo tablet
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dapagliflozin — 10 mg tablet, oral, once daily, 24- week treatment and 80-week extension period
  Arms: 1
Drug: Placebo — matching placebo tablet, oral, once daily, 24- week treatment and 80-week extension period
  Arms: 2

SUMMARY:
This study is carried out to assess whether dapagliflozin improves glycemic control, decreases fasting plasma glucose levels, body weight and blood pressure when added to patient's existing medications and how it compares with their usual treatment without added dapagliflozin. Safety data will be collected and analysed to confirm that treatment with dapagliflozin is safe and well tolerated in patients who have diabetes and cardiovascular disease

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes mellitus.
* Cardiovascular disease
* Uninterrupted anti-diabetic treatment for at least 8 weeks before enrolment

Exclusion Criteria:

* Patients with type 1 diabetes or diabetes insipidus
* Patients with 3 or more oral anti-hyperglycaemic drugs with or without insulin and/or poorly controlled diabetes
* Any clinically significant illness, which would compromise the patient's safety and their participation in the study

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 964 (Actual)
Dates: Start 2010-03; Primary Completion 2011-05 (Actual); Study Completion 2012-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr. Lawrence A Leiter, MD, Principal Investigator — Division of Endocrinology & Metabolism, St Michael's Hospital
Locations (135):
- United States (57):
  - Research Site, Birmingham, Alabama
  - Research Site, Scottsdale, Arizona
  - Research Site, Anaheim, California
  - Research Site, Bell Gardens, California
  - Research Site, Chino, California
  - Research Site, Chula Vista, California
  - Research Site, Huntington Beach, California
  - Research Site, Los Angeles, California
  - Research Site, Mission Hills, California
  - Research Site, Redondo Beach, California
  - Research Site, Riverside, California
  - Research Site, Sacramento, California
  - Research Site, San Diego, California
  - Research Site, Torrance, California
  - Research Site, Aventura, Florida
  - Research Site, Boca Raton, Florida
  - Research Site, Bradenton, Florida
  - Research Site, Brooksville, Florida
  - Research Site, Clearwater, Florida
  - Research Site, Dania Beach, Florida
  - Research Site, Delray Beach, Florida
  - Research Site, New Smyrna Beach, Florida
  - Research Site, Orlando, Florida
  - Research Site, Springfield, Illinois
  - Research Site, Avon, Indiana
  - Research Site, Franklin, Indiana
  - Research Site, Greenfield, Indiana
  - Research Site, Muncie, Indiana
  - Research Site, Waterloo, Iowa
  - Research Site, Topeka, Kansas
  - Research Site, Paducah, Kentucky
  - Research Site, Alexandria, Louisiana
  - Research Site, Rockville, Maryland
  - Research Site, Kalamazoo, Michigan
  - Research Site, Livonia, Michigan
  - Research Site, Billings, Montana
  - Research Site, Berlin, New Jersey
  - Research Site, Brick, New Jersey
  - Research Site, Asheboro, North Carolina
  - Research Site, Fargo, North Dakota
  - Research Site, Cincinnati, Ohio
  - Research Site, Oklahoma City, Oklahoma
  - Research Site, Altoona, Pennsylvania
  - Research Site, Erie, Pennsylvania
  - Research Site, Holland, Pennsylvania
  - Research Site, Lancaster, Pennsylvania
  - Research Site, Media, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Austin, Texas
  - Research Site, Corpus Christi, Texas
  - Research Site, Dallas, Texas
  - Research Site, Irving, Texas
  - Research Site, Richardson, Texas
  - Research Site, San Antonio, Texas
  - Research Site, Sugarland, Texas
  - Research Site, Alexandria, Virginia
  - Research Site, Manassas, Virginia
- Argentina (5):
  - Research Site, Buenos Aires, Buenos Aires F.D.
  - Research Site, Córdoba, Córdoba Province
  - Research Site, Salta, Salta Province
  - Research Site, Rosario, Santa Fe Province
  - Research Site, Santa Fe, Santa Fe Province
- Australia (12):
  - Research Site, Blacktown, New South Wales
  - Research Site, Broadmeadow, New South Wales
  - Research Site, Hornsby, New South Wales
  - Research Site, Wollongong, New South Wales
  - Research Site, Carina Heights, Queensland
  - Research Site, Kippa-Ring, Queensland
  - Research Site, Adelaide, South Australia
  - Research Site, Bedford Park, South Australia
  - Research Site, Keswick, South Australia
  - Research Site, Box Hill, Victoria
  - Research Site, Heidelberg, Victoria
  - Research Site, Herston
- Research Site, Vienna, Austria
- Bulgaria (8):
  - Research Site, Blagoevgrad
  - Research Site, Pernik
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sevlievo
  - Research Site, Sofia
  - Research Site, Stara Zagora
  - Research Site, Varna
- Canada (12):
  - Research Site, Calgary, Alberta
  - Research Site, Edmonton, Alberta
  - Research Site, Moncton, New Brunswick
  - Research Site, Bay Roberts, Newfoundland and Labrador
  - Research Site, Halifax, Nova Scotia
  - Research Site, Etobicoke, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Scarborough Village, Ontario
  - Research Site, Thornhill, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Mirabel, Quebec
  - Research Site, Québec, Quebec
- Research Site, Santiago, Santiago Metropolitan, Chile
- Germany (5):
  - Research Site, Damme
  - Research Site, Dortmund
  - Research Site, Homburg
  - Research Site, Münster
  - Research Site, Wangen
- Hungary (9):
  - Research Site, Ajka
  - Research Site, Balatonfüred
  - Research Site, Budapest
  - Research Site, Esztergom
  - Research Site, Győr
  - Research Site, Komárom
  - Research Site, Mosonmagyaróvár
  - Research Site, Tát
  - Research Site, Veszprém
- Poland (25):
  - Research Site, Bialystok
  - Research Site, Chrzanów
  - Research Site, Gdansk
  - Research Site, Grodzisk Mazowiecki
  - Research Site, Iława
  - Research Site, Kielce
  - Research Site, Krakow
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Mrągowo
  - Research Site, Nowy Sącz
  - Research Site, Poznan
  - Research Site, Płock
  - Research Site, Ruda Śląska
  - Research Site, Skierniewice
  - Research Site, Sopot
  - Research Site, Tarnów
  - Research Site, Torun
  - Research Site, Warsaw
  - Research Site, Wroclaw
  - Research Site, Zabrze
  - Research Site, Zgierz
  - Research Site, Zielona Góra
  - Research Site, Łęczna
  - Research Site, Łęczyca

REFERENCES:
- [Derived] Natale P, Tunnicliffe DJ, Toyama T, Palmer SC, Saglimbene VM, Ruospo M, Gargano L, Stallone G, Gesualdo L, Strippoli GF. Sodium-glucose co-transporter protein 2 (SGLT2) inhibitors for people with chronic kidney disease and diabetes. Cochrane Database Syst Rev. 2024 May 21;5(5):CD015588. doi: 10.1002/14651858.CD015588.pub2. PMID 38770818

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First participant enrolled 15 Mar 2010, last part. last visit for 24-week period: 30 May 2011. 1489 part. enrolled, 964 randomized in USA, Canada, Australia, Chile, Argentina and 5 European countries (value presented in 'Enrolment' field). One add. part. treated but not randomized. Part. with T2DM and CVD who showed inadequate glycemic control.
Pre-assignment Details: During a placebo lead-in period, participants were counselled on dietary and life-style modifications. Anti-diabetic therapy should be kept constant 4 weeks prior to enrolment. Participants eligible for the study were stratified according to age (<65 years or ≥65 years), insulin use and time from most recent qualifying CV event (>1 or ≤1 year).
Groups:
- Dapagliflozin: Dapagliflozin 10 mg plus usual care
- Placebo: Placebo plus usual care
Period: Overall Study
Arm/Group | Dapagliflozin | Placebo
Started | 482 (Of 482 part. 480 were included in full analysis set. Thereof, 1 part. treated but not randomized.) | 483 (Of the 483 participants only 482 were included in the full analysis set.)
Completed | 441 | 428
Not Completed | 41 | 55
Not completed — Adverse Event | 4 | 12
Not completed — Death | 2 | 1
Not completed — Withdrawal by Subject | 8 | 16
Not completed — Lost to Follow-up | 0 | 2
Not completed — Poor/non-compliance | 3 | 4
Not completed — Subject no longer meets study criteria | 15 | 13
Not completed — Incorrect enrollment | 6 | 4
Not completed — Safety | 0 | 2
Not completed — Administrative reason by sponsor | 0 | 1
Not completed — Various | 3 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set defined as all randomized participants (as randomized) who received at least one dose of double-blind study medication, who have a non-missing baseline value and at least one post-baseline efficacy value for at least one efficacy variable during double-blind treatment period.
Groups:
- Total: Total of all reporting groups
Arm/Group | Dapagliflozin | Placebo | Total
Number analyzed (Participants) | 480 | 482 | 962
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.9 (7.60) | 63.6 (7.02) | 63.8 (7.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 159 | 159 | 318
  Male | 321 | 323 | 644
Race/Ethnicity, Customized [Number; unit: Participants]
  White | 454 | 449 | 903
  Black/African American | 9 | 10 | 19
  Asian | 6 | 7 | 13
  Other | 11 | 16 | 27
HbA1c [Mean (Standard Deviation); unit: Percent] | 8.04 (0.759) | 8.08 (0.795) | 8.06 (0.777)
Body weight [Mean (Standard Deviation); unit: kg] | 94.53 (17.804) | 93.23 (16.842) | 93.88 (17.332)
Systolic Blood Pressure [Mean (Standard Deviation); unit: mmHg] | 134.9 (14.53) | 134.6 (13.96) | 134.7 (14.24)
Number of participants with BMI >= 27 kg/m2 at baseline [Number; unit: Participants]
  < 25 kg/m² | 15 | 31 | 46
  >= 25 kg/m² | 465 | 451 | 916
  >= 27 kg/m² | 428 | 416 | 844
  >= 30 kg/m² | 339 | 325 | 664

OUTCOME MEASURES:

1. Primary Outcome: Adjusted Mean Change in HbA1c Levels
Description: To compare the glycemic efficacy of dapagliflozin 10 mg versus placebo when added to usual care in type 2 diabetes patients with cardiovascular disease, measured as the mean change in HbA1c from baseline to week 24.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, participants with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 474 | 471
Percent | -0.33 (0.0434) [-0.42 to -0.25] | 0.07 [-0.02 to 0.15]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.025 (2-sided). A hierarchical closed testing procedure was used to control Type I error across the primary & key secondary objectives; with treatment group and stratum as effects and baseline value as covariate for each endpoint; Mean Difference (Final Values) = -0.40, 95% CI 2-sided [-0.50 to -0.30], Standard Error of Mean 0.0489 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

2. Primary Outcome: Proportion of Responders Meeting All Criteria of a 3-item Endpoint of Clinical Benefit
Description: To compare the clinical benefit of dapagliflozin 10 mg versus placebo when added to usual care in type 2 diabetes patients with cardiovascular disease at week 24, measured as the proportion of responders for a 3-item endpoint of clinical benefit, defined as an absolute drop of 0.5% or more from baseline HbA1c, and a relative drop of 3% or more from baseline for total body weight, and an absolute drop of 3 mmHg or more from baseline in seated systolic blood pressure.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, subjects with non-missing baseline and Week 24 (LOCF) values
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 468 | 469
Percentage of participants | 10.0 (0.7) [7.3 to 12.8] | 1.9 (7.3) [0.7 to 3.2]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: proportion(treat) minus proportion(placebo) = 0 versus the alternative HA: proportion(treat) minus proportion(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel — [p-value comment as in outcome 1, analysis 1]; with age-by-insulin use-by-time from most recent qualifying CV event as stratum; Risk Difference (RD) = 7.0, 95% CI 2-sided [4.3 to 9.8]

3. Secondary Outcome: Adjusted Mean Percent Change in Body Weight
Description: To compare the mean percent change in body weight from baseline to week 24 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, subjects with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of Body Weight
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 480 | 481
Percentage of Body Weight | -2.53 (0.1770) [-2.87 to -2.18] | -0.61 (0.1736) [-0.96 to -0.26]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significant at alpha=0.05 (2-sided). Primary and key secondary endpoints are tested following a hierarchical closed testing procedure; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -1.93, 95% CI 2-sided [-2.31 to -1.54], Standard Error of Mean 0.1957 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

4. Secondary Outcome: Proportion of Participants With a Reduction From Baseline of 5% or More in Body Weight in Participants With Baseline BMI ≥27 kg/m²
Description: To compare the proportion of participants with BMI baseline ≥27 kg/m2 with a reduction from baseline of 5% or more in body weight with dapagliflozin 10 mg versus placebo from baseline to week 24. Least Squares Mean represents the percent of participants adjusted for baseline body weight and age stratum.
Time Frame: Baseline to Week 24
Population: Full Analysis Set, subjects with baseline BMI ≥27 kg/m2 and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 428 | 415
Percentage of participants | 18.4 (1.051) [14.8 to 22.1] | 4.8 (1.876) [2.8 to 6.9]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Superiority or Other; p < 0.0001, Regression, Logistic — [p-value comment as in outcome 3, analysis 1]; Based on methodology of Zhang, Tsiatis & Davidian and Davidian, Tsiatis, Zhang & Lu, with adjustment for baseline total body weight and age stratum; Risk Difference (RD) = 13.6, 95% CI 2-sided [9.4 to 17.8], Standard Error of Mean 2.149

5. Secondary Outcome: Adjusted Mean Change in Systolic Blood Pressure at Week 8 (LOCF)
Description: To compare the mean change in seated systolic blood pressure from baseline to week 8 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 8
Population: Full Analysis Set, subjects with non-missing baseline and Week 8 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 473 | 479
mmHg | -1.85 (0.7105) [-3.25 to -0.45] | 0.86 (0.7135) [-0.53 to 2.26]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0007, ANCOVA — [p-value comment as in outcome 3, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -2.71, 95% CI 2-sided [-4.28 to -1.15], Standard Error of Mean 0.7977 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

6. Secondary Outcome: Adjusted Mean Change in Seated Systolic Blood Pressure at Week 24 (LOCF)
Description: To compare the mean change in seated systolic blood pressure from baseline to week 24 between dapagliflozin 10 mg versus placebo.
Time Frame: Baseline to Week 24
Population: Full Analysis set, subjects with non-missing baseline and Week 24 (LOCF) values
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 473 | 479
mmHg | -2.70 (0.7109) [-4.10 to -1.30] | 0.32 (0.7140) [-1.07 to 1.72]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0002, ANCOVA — [p-value comment as in outcome 3, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -3.02, 95% CI 2-sided [-4.59 to -1.46], Standard Error of Mean 0.7983 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

7. Secondary Outcome: Adjusted Mean Change in Seated Systolic Blood Pressure (SBP) at Week 8 (LOCF) in Participants With Baseline SBP>=130 mmHg
Description: To compare the mean change in seated systolic blood pressure (SBP) in participants with baseline seated SBP ≥130 mmHg achieved with dapagliflozin versus placebo from baseline to week 8.
Time Frame: Baseline to Week 8
Population: Full Analysis set, participants with baseline seated SBP ≥130 mmHg and Week 8 (LOCF) value
Measure: Least Squares Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Dapagliflozin | Placebo
Number analyzed (Participants) | 300 | 309
mmHg | -5.33 (0.8612) [-7.02 to -3.64] | -1.89 (0.8612) [-3.58 to -0.20]
Statistical Analysis 1: Comparison: Dapagliflozin vs Placebo; H0: mean(treat) minus mean(placebo) = 0 versus the alternative HA: mean(treat) minus mean(placebo) =/= 0; Test type: Superiority or Other; p = 0.0004, ANCOVA — [p-value comment as in outcome 3, analysis 1]; with treatment group and stratum as effects and baseline value as covariate; Mean Difference (Final Values) = -3.44, 95% CI 2-sided [-5.35 to -1.53], Standard Error of Mean 0.9746 — with stratum = age-by-insulin use-by-time from most recent qualifying CV event

ADVERSE EVENTS:
Time Frame: Non-serious / serious adverse events on or after the first day and on or prior to the last day of the 24-week double-blind treatment plus 4/30 days or up to follow-up visit if earlier, or up to and including the start date of extension period if earlier.
Description: Participants were questioned at each study visit about the occurrence of any health problems and any examination conducted at a study visit was assessed in comparison to the status at study entry.
Arm/Group | Dapagliflozin | Placebo
Serious Adverse Events (participants affected / at risk) | 41/482 | 46/483
Other Adverse Events (participants affected / at risk) | 147/482 | 134/483
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Dapagliflozin (N=482) | Placebo (N=483)
Angina unstable (Cardiac disorders) | 3 | 2
Myocardial infarction (Cardiac disorders) | 3 | 1
Acute coronary syndrome (Cardiac disorders) | 2 | 0
Atrial fibrillation (Cardiac disorders) | 2 | 3
Angina pectoris (Cardiac disorders) | 1 | 1
Cardiac failure (Cardiac disorders) | 1 | 1
Coronary artery disease (Cardiac disorders) | 1 | 1
Ventricular tachycardia (Cardiac disorders) | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 1
Cardiac failure congestive (Cardiac disorders) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 2 | 0
Dizziness (Nervous system disorders) | 1 | 1
Ischaemic stroke (Nervous system disorders) | 1 | 1
Spinal cord compression (Nervous system disorders) | 1 | 0
Syncope (Nervous system disorders) | 1 | 1
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Respiratory tract infection (Infections and infestations) | 2 | 1
Bronchitis (Infections and infestations) | 1 | 0
Osteomyelitis (Infections and infestations) | 1 | 0
Peritonsillar abscess (Infections and infestations) | 1 | 0
Gastroenterits (Infections and infestations) | 0 | 1
Herpes zoster (Infections and infestations) | 0 | 1
Lung abscess (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 0 | 2
Pyelonephritis (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Meningioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Renal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 0
Gastric polyps (Gastrointestinal disorders) | 1 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 1
Small intestine obstruction (Gastrointestinal disorders) | 0 | 1
Intervertebral disc disorder (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Bladder diverticulum (Renal and urinary disorders) | 1 | 0
Renal failure (Renal and urinary disorders) | 1 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure acute (Renal and urinary disorders) | 0 | 1/482
Peripheral arterial occlusive disease (Vascular disorders) | 2 | 2/482
Diabetic vascular disorder (Vascular disorders) | 1 | 0/482
Circulatory collapse (Vascular disorders) | 0 | 1/482
Deep vein thrombosis (Vascular disorders) | 0 | 1/482
Extremity necrosis (Vascular disorders) | 0 | 1/482
Hypertensive crisis (Vascular disorders) | 0 | 1/482
Peripheral ischaemia (Vascular disorders) | 0 | 1/482
Thrombosis (Vascular disorders) | 0 | 1/482
Angioedema (Skin and subcutaneous tissue disorders) | 1 | 0/482
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0/482
Drug hypersensitivity (Immune system disorders) | 1 | 0/482
Excoriation (Injury, poisoning and procedural complications) | 1 | 0/482
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1/482
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1/482
Contusion (Injury, poisoning and procedural complications) | 0 | 1/482
Femoral neck fracture (Injury, poisoning and procedural complications) | 0 | 1/482
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1/482
Vascular graft thrombosis (Injury, poisoning and procedural complications) | 0 | 1/482
Blood parathyroid hormone decreased (Investigations) | 1 | 0/482
Hypoglycaemia (Metabolism and nutrition disorders) | 1 | 0/482
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 1/482
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1/482
Angioplasty (Surgical and medical procedures) | 1 | 0/482
Acute vestibular syndrome (Ear and labyrinth disorders) | 0 | 1/482
Chest pain (General disorders) | 0 | 3
Schizophrenia, paranoid type (Psychiatric disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Dapagliflozin (N=482) | Placebo (N=483)
Urinary tract infection (Infections and infestations) | 27 | 18
Nasopharyngitis (Infections and infestations) | 26 | 26
Upper respiratory tract infection (Infections and infestations) | 15 | 24
Hypoglycemia (Endocrine disorders) | 101 | 84

LIMITATIONS AND CAVEATS:
For participants who did not complete 8 and/or 24 weeks, respectively, LOCF was used. For HbA1c: excluding data after glycemic rescue, Weight: including data after rescue, SBP: excluding data after anti-hypertensive rescue.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an Investigator requests permission to publish data from this study any such publication is to be agreed with AstraZeneca (AZ) in advance. The investigator agrees to provide AZ as soon as possible with drafts of proposed publications. Unless otherwise agreed, AZ shall have a period of 60 days from receipt of the proposed final manuscript to review it and may within such time require that submission for publication of the manuscript be delayed in order for AZ to file patent applications.